CLINICAL TRIAL: NCT00662194
Title: A Study of Innate Immunity in HIV Positive Patients Co-infected With Hepatitis C or Hepatitis B
Brief Title: Innate Immunity in HIV Positive Patients Co-infected With Hepatitis C Virus (HCV) or Hepatitis B Virus (HBV)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: Monash Medical Centre (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ALF-55/08
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: HIV-hepatitis Co-infection; HIV Infections
Keywords: HIV; HBV; HCV; co-infection; innate immunity
MeSH Terms: conditions — HIV Infections; Coinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- 1: HIV-HBV co-infected and receiving anti-retroviral therapy (ART) and CD4 count > 500cells/mm3
- 2: HIV-HBV co-infected and receiving ART and CD4 count 200-500 cells/mm3
- 3: HIV-HBV co-infected and receiving ART and CD4 count <200cells/mm3
- 4: HIV-HBV co-infected and not receiving ART
- 5: HIV-HCV co-infected & receiving anti-retroviral therapy (ART) and CD4 count > 500cells/mm3
- 6: HIV-HCV co-infected and receiving ART and CD4 count 200-500 cells/mm3
- 7: HIV-HCV co-infected and receiving ART and CD4 count <200cells/mm3
- 8: HIV-HCV co-infected and not receiving ART

SUMMARY:
Data from this study will provide the first information how the innate immune system may be altered in HIV-HCV and HIV-HBV co-infected individuals, and describe Toll-like receptor changes with HIV co-infection therapy.

DETAILED DESCRIPTION:
It has been demonstrated that Toll-like receptors (TLR) are involved in viral hepatitis - hepatitis B (HBV), hepatitis C (HCV) - and HIV in the setting of mono-infection. However the role of innate immunity in the pathogenesis of HIV-hepatitis co-infection in both natural and therapy-associated viral clearance remains unclear. The data from this study may reveal patterns which could predict how and when patients spontaneously, and with therapy, resolve HBV or HCV in the setting of co-infection.

The aim of the study is to evaluate the activity of innate immunity in different subsets of HIV-infected populations co-infected with chronic hepatitis B and/or C. Our hypothesis is that innate immunity is altered in HIV and hepatitis co-infection and that this differs from both hepatitis and HIV mono-infection.

The study is a cross-sectional and longitudinal pilot study of individuals infected with HIV and either HBV or HCV.

ELIGIBILITY:
Inclusion Criteria:

* HIV and either HBV or HCV co-infection
* 18 years and older
* able to give informed consent

Exclusion Criteria:

* HIV-HBV-HCV triple infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
TLR change with HIV co-infection therapy | 6 months

SECONDARY OUTCOMES:
TLR change patterns on spontaneously and on treatment resolved HBV or HCV in the co-infected setting | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joe Sasadeusz, MD, PhD, Principal Investigator — The Alfred
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia